CLINICAL TRIAL: NCT01023048
Title: First Use of Parental Support Technology(R) for Single Gene Analysis Plus Aneuploidy Screening in Preimplantation Genetic Diagnosis
Brief Title: Concurrent Single Gene and 24 Chromosome Aneuploidy Preimplantation Genetic Diagnosis (PGD)
Acronym: IVF008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVF008
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Any Single Gene Disorder (Cystic Fibrosis, Tay-Sachs)
Keywords: preimplantation diagnosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PGD testing (Experimental)
  Interventions: Other: preimplantation diagnosis

INTERVENTIONS:
Other: preimplantation diagnosis — genetic testing on embryos to identify embryos that are affected by a single gene disorder (e.g. cystic fibrosis, Tay-Sachs, sickle cell anemia)
  Other Names: Parental Support Technology

SUMMARY:
Gene Security Network has developed a novel technology called Parental SupportTM (PS) which is used for Preimplantation Genetic Screening/Diagnosis (PGS/D) during in vitro fertilization (IVF). This technology allows IVF physicians to identify embryos, prior to transfer to the uterus, which have the best chance of developing into healthy children. The purpose of this study is to validate clinical use of PS to detect specific genetic mutation(s) known to cause severe inheritable diseases in embryos produced by at-risk couples. This may be done while simultaneously testing these embryos for aneuploidy. This study will allow for first of its kind commercial PGS/D testing to detect disease-associated genetic mutations together with aneuploidy screening.

ELIGIBILITY:
Inclusion Criteria:

* couple (mother and father)at risk to have a child with a single gene disorder (e.g. cystic fibrosis, Tay-Sachs, sickle cell anemia)
* Able to provide laboratory report from commercial CLIA certified laboratory confirming presence of disease associated mutation in mother and/or father
* couple planning to go through IVF and desiring PGD for the specified mutation
* Father (male) willing and able to provide sperm sample
* Maternal (female's) age <40 years (e.g., 39 or younger)
* CVS/Amnio planned once the pregnancy occurs; willing/able to provide amnio/cvs sample for confirmatory testing or provide test results of confirmatory testing performed by an external CLIA certified laboratory.
* FSH <10 (FSH = Follicle Stimulating Hormone. FSH is an indicator of egg quality and rough predictor of egg stimulation success. FSH is routinely measured by the IVF center prior to beginning an IVF cycle.)

Exclusion Criteria:

* Couples without prior documentation of genetic mutation as specified above
* Adult couples where the male partner is not willing, able, or available to provide a semen sample.
* Maternal age >=40 years
* Couple unwilling to have amnio/cvs

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2009-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Confirm diagnosis through prenatal diagnosis (CVS or amniocentesis) | 10-20 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rabinowitz, PhD, Principal Investigator — Natera, Inc.
Locations (1):
- Gene Security Network, Redwood City, California, United States